CLINICAL TRIAL: NCT00118040
Title: Phase II Study of Isoflavone G-2535 (Genistein) in Patients With Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2013-00453; NCI-2013-00453 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000433520; WCCC-UWI03-1-01; WCCC-CO-04307; UWI03-1-01 (Other: University of Wisconsin Chemoprevention Consortium); UWI03-1-01 (Other: DCP); N01CN35153 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-03

CONDITIONS: Recurrent Bladder Carcinoma; Stage I Bladder Cancer AJCC v6 and v7; Stage II Bladder Cancer AJCC v6 and v7; Stage III Bladder Cancer AJCC v6 and v7
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm I (lower dose genistein) (Experimental): Patients receive oral genistein twice daily for approximately 14-30 days. One day after completion of genistein or placebo, all patients undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.
  Interventions: Drug: Genistein; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery
- Arm II (higher dose genistein) (Experimental): Patients receive oral genistein as in arm I but at a higher dose. One day after completion of genistein or placebo, all patients undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.
  Interventions: Drug: Genistein; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery
- Arm III (placebo) (Placebo Comparator): Patients receive oral placebo twice daily for approximately 14-30 days. One day after completion of genistein or placebo, all patients undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo Administration; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Genistein — Given orally
  Other Names: 4'',5, 7-Trihydroxyisoflavone; Genestein; Genisteol; Prunetol
  Arms: Arm I (lower dose genistein); Arm II (higher dose genistein)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo Administration — Given orally
  Arms: Arm III (placebo)
Procedure: Therapeutic Conventional Surgery — Undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.

SUMMARY:
Studying samples of blood, urine, and tissue from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer. It may also help doctors learn how genistein or placebo works in patients with bladder cancer. This randomized phase II trial is studying genistein or placebo to compare how they work in patients who are undergoing surgery for bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure the effect of G-2535 on EGF-R phosphorylation. Two EGF-R phosphorylation sites with functional significance are phosphotyrosine 992, which is a direct binding site for the PLC-gamma SH2 domain, and phosphotyrosine 1068, a binding site for the Grb2/SH2 domain. The expression of EGF-R and phosphorylated EGF-R will be determined in tumors as well as adjacent and remote normal appearing urothelium.

SECONDARY OBJECTIVES:

I. Measuring tissue intermediate endpoint biomarkers such as EGF-R mutations (EGFR vIII, exon 19-21), Ki67, activated Caspase 3, Akt, P-Akt, MAP kinase, P-MAP kinase, COX-2, survivin, and BLCA-4 and we will also determine survivin and BLCA-4 levels in urine specimens as surrogate tumor markers. Biomarkers associated with the EGF-R pathway, including Akt and P-Akt will be studied by immunohistochemistry. Additionally, Ki67, activated Caspase 3 (as a marker of apoptosis), and COX-2 will serve as biological endpoint biomarkers to measure the effects of G-2535 on proliferation, apoptosis, and other processes and molecules relevant to bladder cancer. These studies will be performed on tumors as well as adjacent and remote normal urothelium. II. Safety will also be studied.

OUTLINE: This is a randomized, placebo-controlled, multicenter study. Patients are stratified according to invasiveness of disease (non-invasive [stage Ta, Tis, or T1] vs invasive [stage T2, T3, or T4]). Patients are randomized to 1 of 3 treatment arms.

Arm I: Patients receive oral genistein twice daily for approximately 14-30 days.

Arm II: Patients receive oral genistein as in arm I but at a higher dose. Arm III: Patients receive oral placebo twice daily for approximately 14-30 days.

One day after completion of genistein or placebo, all patients undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.

Patients undergo blood, urine, and tissue sample collection for pharmacogenomic, pharmacokinetic, and biomarker laboratory studies. Blood and urine samples are collected at baseline, after 1 week of treatment, and at the time of surgery for pharmacokinetic and urine biomarker (survivin and BLCA-4) studies. Pharmacogenomic studies (epidermal growth factor receptor [EGFR] polymorphisms and CYP3A 4/5 genotypes) are performed at baseline using blood samples. Tissue biomarker (EGFR polymorphism, EGFR mutations [EGFR vIII, exon 19-21], EGFR, phosphorylated EGFR, Ki67, activated caspase 3, Akt, P-Akt, MAP kinase, P-MAP kinase, COX-2, survivin, and BLCA4) studies using tumor tissue and adjacent and remote normal urothelium are performed at baseline and at the completion of treatment.

PROJECTED ACCRUAL: A total of 60 patients (20 per treatment arm) will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for this study will have been evaluated by diagnostic office cystoscopy and found to have a bladder tumor; enrollment (signing of the consent form) must be within 60 days of pre-study cystoscopy demonstrating bladder tumor; the participant should have no evidence of distant metastasis and the primary tumor may represent either an initial diagnosis or recurrent disease of any clinical stage. Study participants must also be candidates for either subsequent cystoscopy/transurethral resection of bladder tumor (TURBT) or complete or partical cystectomy; histologic diagnosis is not required for enrollment; pre-enrollment diagnostic cystoscopy must be at least 45 days after treatment of the bladder with other agents such as BCG (participants with recurrent disease)
* ECOG performance status 0 or 1
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document
* WBC >= 3000/mm^3
* Platelets >= 100,000mm^3
* Hemoglobin >= 10 g/dL
* Bilirubin =< 1.4 mg/dl
* AST =< 3x normal
* Creatinine =< 2.0mg/dl
* Serum calcium =< 10.2 mg/dl,
* Amylase =< 3 x normal
* Na >= 125 and =< 155 mmol/L
* K >= 3.2 and =< 6 mmol/L
* Cl >= 85 and =< 114 mmol/L
* CO2 >= 11 mEQ/dL
* TSH within 1.3 x the upper range of normal and normal T4
* Females of child-bearing potential must have a negative pregnancy test; patients who have had a bilateral oophorectomy, hysterectomy, are greater than 1 year since their last menses, or are greater than 51 years of age are not considered to be of child-baring potential
* Participants must agree to stop soy supplements before enrolling in the study
* Patients must agree to stop taking NSAIDS before enrolling in the study; patients may, however, take cardioprotective doses of aspirin equal to or less than 81mg per day

Exclusion Criteria:

* Participant may not have received other treatment for bladder cancer between the pre-enrollment cystoscopy and subsequent surgery
* Participants may not be receiving any other investigational agents
* Participant may not have received prior pelvic irradiation for any reason
* Participant may not be receiving concurrent systemic cancer treatment for other cancers
* Participant may not be taking concurrent soy supplements while on the study medication
* Participant may not be taking concurrent NSAIDS (aspirin doses of =< 81 mg acceptable) while on the study medication
* Participant may not be taking thyroid medications
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to genistein, soy isoflavones or other allergies to soy-based products will render a participant ineligible
* Uncontrolled concurrent illness will render a participant ineligible including, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unregulated cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women may not be pregnant or lactating; the effects of G-2535 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-06-24 (Actual); Primary Completion 2010-08-15 (Actual); Study Completion 2010-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard H Bailey, Principal Investigator — University of Wisconsin Chemoprevention Consortium
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - South Orange County Surgical Medical Group Inc, Laguna Hills, California
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - AccuMed Research Associates, Garden City, New York
  - University of Rochester, Rochester, New York
  - Urology San Antonio Research PA, San Antonio, Texas
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Chemoprevention Consortium, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin

REFERENCES:
- [Derived] Messing E, Gee JR, Saltzstein DR, Kim K, diSant'Agnese A, Kolesar J, Harris L, Faerber A, Havighurst T, Young JM, Efros M, Getzenberg RH, Wheeler MA, Tangrea J, Parnes H, House M, Busby JE, Hohl R, Bailey H. A phase 2 cancer chemoprevention biomarker trial of isoflavone G-2535 (genistein) in presurgical bladder cancer patients. Cancer Prev Res (Phila). 2012 Apr;5(4):621-30. doi: 10.1158/1940-6207.CAPR-11-0455. Epub 2012 Jan 31. PMID 22293631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited during a 3 year period by staff at 7 participating institutions (both University hospitals and community clinics).
Groups:
- Arm I (300mg Genistein): Patients receive oral genistein (150mg) twice daily for approximately 14-30 days. One day after completion of genistein or placebo, all patients undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.
- Arm II (600mg Genistein): Patients receive oral genistein as in arm I but at a higher dose (600mg). One day after completion of genistein or placebo, all patients undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.
Period: Overall Study
Arm/Group | Arm I (300mg Genistein) | Arm II (600mg Genistein) | Arm III (Placebo)
Started | 20 | 20 | 20
Completed | 19 | 18 | 14
Not Completed | 1 | 2 | 6
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Medical Contraindication | 0 | 0 | 1
Not completed — Non-Compliant Participant | 1 | 1 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (300mg Genistein) | Arm II (600mg Genistein) | Arm III (Placebo) | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 7 | 22
  >=65 years | 12 | 13 | 13 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.60 (9.16) | 68.65 (9.16) | 71.95 (12.67) | 69.73 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 2 | 8
  Male | 15 | 19 | 18 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 20 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 20 | 20 | 20 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Epidermal Growth Factor Receptor (EGFR) Phosphorylation in Tumor Tissue, as Measured by Immunohistochemistry After the Completion of Treatment
Description: Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days
Population: For this outcome Arm 1 and Arm II were analyzed together which lead to Arm IV. Also for Arm III although 14 participants successfully completed the study for this group they were able to analyzed 15 for this outcome.
Measure: Number; unit: percentage of pEGFR strength signal
Groups:
- Arm IV (300mg Genistein + 600mg Genistein): This is a combination analysis those on 300mg of genistein and 600mg genistein
Arm/Group | Arm I (300mg Genistein) | Arm II (600mg Genistein) | Arm III (Placebo) | Arm IV (300mg Genistein + 600mg Genistein)
Number analyzed (Participants) | 19 | 18 | 15 | 37
percentage of pEGFR strength signal
  Strong | 52.63 | 83.33 | 93.33 | 67.57
  Moderate | 21.35 | 16.67 | 0.00 | 18.92
  Weak | 26.32 | 0.00 | 6.67 | 13.51
  Negative | 0.00 | 0.00 | 0.00 | 0.00

2. Secondary Outcome: BLCA-4 in Urine by Visit
Description: Detecting the mean amount of the biomarker BLCA-4 in the urine of patients prior to starting study agent, at Day 8 and pre-surgery time (when they have been on study agent between 14-21 days). This is measured by urine analysis at each of the time points to serve as a surrogate tumor marker.
Time Frame: up to 21 days
Population: For this outcome Arm 1 and Arm II were analyzed together which lead to Arm IV. Also for Arm III although 14 participants successfully completed the study for this group they were able to analyzed 17 for this outcome.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 39 | 17 | 20 | 19
pg/ml
  Baseline | 0.54 (0.35) | 0.46 (0.24) | 0.52 (0.37) | 0.55 (0.34)
  Day 8 | 0.52 (0.42) | 0.53 (0.20) | 0.54 (0.42) | 0.50 (0.43)
  Pre-Surgery | 0.52 (0.36) | 0.49 (0.34) | 0.59 (0.39) | 0.44 (0.31)

3. Secondary Outcome: Survivin in Urine by Visit (pg/ml)
Description: Detecting the mean amount of the biomarker Survivin in the urine of patients prior to starting study agent, at Day 8 and pre-surgery time (when they have been on study agent between 14-21 days). This is measured by urine analysis at each of the time points to serve as a surrogate tumor marker.
Time Frame: up to 21 days
Population: For this outcome Arm 1 and Arm II were analyzed together which lead to Arm IV. Also for Arm III although 14 participants successfully completed the study for this group they were able to analyzed 16 for this outcome.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 16 | 18 | 19
pg/ml
  Baseline | 58.5 (141.3) | 16.0 (37.4) | 71.0 (171.7) | 46.6 (108.6)
  Day 8 | 41.0 (123.8) | 17.8 (32.6) | 60.3 (175.7) | 23.7 (41.1)
  Pre-Surgery | 55.4 (166.7) | 28.6 (43.3) | 84.4 (237.3) | 29.5 (49.6)

4. Secondary Outcome: Survivin in Tumor Tissue
Description: Detecting the signal of the biomarker, Survivin, in the tumor tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of Survivin strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of Survivin strength signal
  Strong | 24.32 | 0.00 | 15.79 | 33.33
  Moderate | 13.51 | 33.33 | 15.79 | 11.11
  Weak | 35.14 | 33.33 | 26.32 | 44.44
  Negative | 27.03 | 33.33 | 42.11 | 11.11

5. Secondary Outcome: EGFR Mutations in Tumor Tissue
Description: Detecting the signal of EGFR mutations in the tumor tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of EGFR strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of EGFR strength signal
  Strong | 48.65 | 46.67 | 42.11 | 55.56
  Moderate | 16.22 | 0.00 | 10.53 | 22.22
  Weak | 16.22 | 6.67 | 21.05 | 11.11
  Negative | 18.92 | 46.67 | 26.32 | 11.11

6. Primary Outcome: pEGFR in Benign Tissue
Description: Detecting the signal of the biomarker, pEGFR, in the benign tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: For this outcome Arm 1 and Arm II were analyzed together which lead to Arm IV.
Measure: Number; unit: percentage of pEGFR strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 22 | 9 | 14 | 8
percentage of pEGFR strength signal
  Strong | 4.55 | 0.00 | 7.14 | 0.00
  Moderate | 27.27 | 33.33 | 28.57 | 25.00
  Weak | 54.55 | 44.44 | 57.14 | 50.00
  Negative | 13.64 | 22.22 | 7.14 | 25.00

7. Secondary Outcome: EGFR in Benign Tissue
Description: Detecting the signal of the biomarker, EGFR, in the benign tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: For this outcome Arm 1 and Arm II were analyzed together which lead to Arm IV.
Measure: Number; unit: percentage of EGFR strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 22 | 9 | 14 | 8
percentage of EGFR strength signal
  Strong | 40.91 | 11.11 | 42.86 | 37.50
  Moderate | 13.64 | 22.22 | 7.14 | 25.00
  Weak | 9.09 | 0.00 | 14.29 | 0.00
  Negative | 36.36 | 66.67 | 35.71 | 37.50

8. Secondary Outcome: Ki-67 in Tumor Tissue
Description: Detecting the signal of the biomarker, Ki-67, in the tumor tissue after being on study drug for between 14-21 days as a way to measuring the effects G-2535 have on it with regards to proliferation, apoptosis, and other processes relevant to bladder cancer.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of Ki-67 strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of Ki-67 strength signal
  Strong | 40.54 | 26.67 | 47.37 | 33.33
  Moderate | 18.92 | 20.00 | 15.79 | 22.22
  Weak | 35.14 | 46.67 | 31.58 | 38.89
  Negative | 5.41 | 6.67 | 5.26 | 5.56

9. Secondary Outcome: Activated Caspase 3 in Tumor Tissue
Description: Detecting the signal of the biomarker, Activated Caspase 3, in the tumor tissue after being on study drug for between 14-21 days as a way to measuring the effects G-2535 have on it with regards to proliferation, apoptosis, and other processes relevant to bladder cancer.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of Caspase 3 strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of Caspase 3 strength signal
  Strong | 10.81 | 0.00 | 10.53 | 11.11
  Moderate | 2.70 | 6.67 | 0.00 | 5.56
  Weak | 27.03 | 26.67 | 26.32 | 27.78
  Negative | 59.46 | 66.67 | 63.16 | 55.56

10. Secondary Outcome: COX2 in Tumor Tissue
Description: Detecting the signal of the biomarker, COX2, in the tumor tissue after being on study drug for between 14-21 days as a way to measuring the effects G-2535 have on it with regards to proliferation, apoptosis, and other processes relevant to bladder cancer.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of COX2 strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of COX2 strength signal
  Strong | 13.51 | 0.00 | 15.79 | 11.11
  Moderate | 32.43 | 26.67 | 36.84 | 27.78
  Weak | 16.22 | 33.33 | 5.26 | 27.78
  Negative | 37.84 | 40.00 | 42.11 | 33.33

11. Secondary Outcome: AKT in Tumor Tissue
Description: Detecting the signal of the biomarker, AKT, in the tumor tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of AKT strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of AKT strength signal
  Strong | 64.86 | 60.00 | 78.95 | 50.00
  Moderate | 10.81 | 13.33 | 5.26 | 16.67
  Weak | 18.92 | 20.00 | 10.53 | 27.78
  Negative | 5.41 | 6.67 | 5.26 | 5.56

12. Secondary Outcome: pAKT in Tumor Tissue
Description: Detecting the signal of the biomarker, pAKT, in the tumor tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of pAKT strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of pAKT strength signal
  Strong | 43.24 | 33.33 | 47.37 | 38.89
  Moderate | 8.11 | 0.00 | 5.26 | 11.11
  Weak | 2.70 | 6.67 | 0.00 | 5.56
  Negative | 45.95 | 60.00 | 47.37 | 44.44

13. Secondary Outcome: MAP Kinase in Tumor Tissue
Description: Detecting the signal of the biomarker, MAP Kinase, in the tumor tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of MAP Kinase strength signal
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of MAP Kinase strength signal
  Strong | 75.68 | 86.67 | 84.21 | 66.67
  Moderate | 16.22 | 6.67 | 10.53 | 22.22
  Weak | 2.70 | 0.00 | 0.00 | 5.56
  Negative | 5.41 | 6.67 | 5.26 | 5.56

14. Secondary Outcome: pMAP Kinase in Tumor Tissue
Description: Detecting the signal of the biomarker, pMAP Kinase, in the tumor tissue after being on study drug for between 14-21 days.
  Strong, Moderate, Weak, and Negative are categorized based on the signal. The measurements display the strength of the signal between the different Arms.
Time Frame: up to 21 days on Study Drug
Population: as for outcome 1
Measure: Number; unit: percentage of pMAP Kinase strength signa
Arm/Group | Arm IV (300mg Genistein + 600mg Genistein) | Arm III (Placebo) | Arm I (300mg Genistein) | Arm II (600mg Genistein)
Number analyzed (Participants) | 37 | 15 | 19 | 18
percentage of pMAP Kinase strength signa
  Strong | 48.65 | 66.67 | 36.84 | 61.11
  Moderate | 37.84 | 20.00 | 42.11 | 33.33
  Weak | 13.51 | 6.67 | 21.05 | 5.56
  Negative | 0.00 | 6.67 | 0.00 | 0.00

ADVERSE EVENTS:
Time Frame: up to 30 days from randomization
Groups:
- Arm III (Placebo): Patients receive oral placebo twice daily for approximately 14-30 days. One day after completion of genistein or placebo, all patients undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.
  laboratory biomarker analysis: Correlative studies
  placebo: Given orally
  therapeutic conventional surgery: Undergo cystoscopic excision, transurethral resection of the bladder tumor, or cystectomy.
  pharmacological study: Correlative studies
Arm/Group | Arm I (Lower Dose Genistein) | Arm II (Higher Dose Genistein) | Arm III (Placebo)
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 18/20 | 17/20 | 12/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lower Dose Genistein) (N=20) | Arm II (Higher Dose Genistein) (N=20) | Arm III (Placebo) (N=20)
Supraventricular arrhythmia- Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lower Dose Genistein) (N=20) | Arm II (Higher Dose Genistein) (N=20) | Arm III (Placebo) (N=20)
Fatigue (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Sweating (Social circumstances) | 0 (0) | 0 (0) | 1 (1)
Itiching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infection of brochus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection of upper airway (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection of urinary tract (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
amylase (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (4)
Bicarbonate, serum low (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Elevated Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
decreased bilirubin (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
decreased bun (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated bun (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1)
Elevated Chloride (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
High chloride (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
hypoatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
lipase (Metabolism and nutrition disorders) | 6 (6) | 1 (1) | 2 (2)
low chloride (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
low creatinine (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
low protein in blood work (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Low total bilirubin (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fullness in left jaw area (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
muscle weakness extremity-upper (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
pain: Breast (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain: Esophagus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain: Muscle (General disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
excess phlegm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
lupus (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
rhinitis (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
decreased red blood cells (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
elevated hematocrit (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
elevated platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
elevated white blood cells (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
high platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
hemoglobin (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 2 (2)
leukocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
low hematocrit (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less